CLINICAL TRIAL: NCT06346392
Title: A Phase III Multi-center, Open-label, Sponsor-blinded, Randomized Study of AZD0901 Monotherapy Compared With Investigator's Choice of Therapy in Second- or Later-Line Adult Participants With Advanced/Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma Expressing Claudin18.2 (CLARITY Gastric 01)
Brief Title: AZD0901 Compared With Investigator's Choice of Therapy in Participants With Second- or Later-line Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma Expressing Claudin18.2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D9802C00001; 2023-508276-11-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-02-28; First posted 2024-04-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
Keywords: Gastric cancer; Gastroesophageal junction cancer; Phase III; Claudin 18.2; AZD0901
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Docetaxel; Irinotecan; trifluridine tipiracil drug combination; apatinib

STUDY DESIGN:
Intervention Model Description: Participants were randomized in a 1:1:1 ratio to one of the following intervention arms until the dose selection decision was made. Randomization will continue in a 1:1 ratio to the 2 remaining arms:
  Arm 1: AZD0901 arm 1 IV, Q3W Arm 2: AZD0901 arm 2 IV, Q3W (Enrolment was closed) Arm 3: Participants in the Investigator's choice arm, including regionally accepted chemotherapies or targeted therapies 2L: Ramucirumab 8 mg/kg IV on Days 1 and 15 and paclitaxel 80 mg/m2 IV on Days 1, 8, and 15, Q4W 2L: Paclitaxel 80 mg/m2 IV on Days 1, 8, and 15, Q4W (for participants with contraindication to ramucirumab only) 2L: Docetaxel 75-100 mg/m2 IV on Day 1, Q3W (for participants with contraindication to ramucirumab only) 3L+: Irinotecan 150-180 mg/m2 IV on Days 1 and 15, Q4W 3L+: TAS-102 35 mg/m2 up to a maximum of 80 mg orally twice a day on Days 1 to 5 and Days 8 to 12, Q4W (except China) 3L+: Apatinib 500-850 mg, orally once daily, Q4W (China only)
Who Masked: Outcomes Assessor
Masking Description: This is an open-label study; however, it will be conducted 'sponsor-blind' and the specific treatment to be taken by a participant will be assigned using an IRT/RTSM. To maintain the integrity of the study, sponsor access to treatment records will be restricted, and, in particular, under no circumstances will the sponsor undertake any efficacy analysis by treatment arm during the study. A Study Integrity Plan will be generated in which nominated individuals who will be granted access to any treatment-revealing data will be pre-specified, with their reason for requiring access detailed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AZD0901 arm 1 (Experimental): Participants in the AZD0901 arm 1 will receive AZD0901 dose level 1 intravenous infusion treatment.
  Interventions: Drug: AZD0901
- AZD0901 Arm 2 (Experimental): Participants in the AZD0901 arm 2 will receive AZD0901 dose level 2 intravenous infusion treatment. (Enrolment was closed)
  Interventions: Drug: AZD0901
- Investigator's choice arm (Active Comparator): Participants in the Investigator's choice arm will receive a regimen of Investigator's choice, including regionally accepted chemotherapies or targeted therapies.
  Interventions: Drug: Ramucirumab+ paclitaxel; Drug: Paclitaxel; Drug: Docetaxel; Drug: Irinotecan; Drug: TAS-102; Drug: Apatinib

INTERVENTIONS:
Drug: AZD0901 — Participants in the AZD0901 arm 1 will receive dose level 1 AZD0901 IV
  Other Names: Sonesitatug Vedotin
  Arms: AZD0901 arm 1
Drug: AZD0901 — Participants in the AZD0901 arm 2 will receive dose level 2 AZD0901 IV (Enrolment was closed)
  Other Names: Sonesitatug Vedotin
  Arms: AZD0901 Arm 2
Drug: Ramucirumab+ paclitaxel — Ramucirumab 8 mg/kg IV on Days 1 and 15 and paclitaxel 80 mg/m2 IV on Days 1, 8, and 15, Q4W
  Arms: Investigator's choice arm
Drug: Paclitaxel — Paclitaxel 80 mg/m2 IV on Days 1, 8, and 15, Q4W (for participants with contraindication to ramucirumab only)
  Arms: Investigator's choice arm
Drug: Docetaxel — Docetaxel 75-100 mg/m2 IV on Day 1, Q3W (for participants with contraindication to ramucirumab only)
  Arms: Investigator's choice arm
Drug: Irinotecan — Irinotecan 150-180 mg/m2 IV on Days 1 and 15, Q4W
  Arms: Investigator's choice arm
Drug: TAS-102 — TAS-102 35 mg/m2 up to a maximum of 80 mg orally twice a day on Days 1 to 5 and Days 8 to 12, Q4W (except China)
  Arms: Investigator's choice arm
Drug: Apatinib — Apatinib 500-850 mg at Investigator's discretion based on participant's condition and tolerability, orally once daily, Q4W (China only)
  Arms: Investigator's choice arm

SUMMARY:
The purpose of this study is to measure the efficacy and safety of AZD0901 compared to Investigator's choice of therapy as 2L+ treatment for participants with advanced or metastatic gastric or GEJ adenocarcinoma expressing CLDN18.2.

DETAILED DESCRIPTION:
This is a Phase III, multi-center, open-label, sponsor-blinded, randomized, global study to assess the efficacy and safety of AZD0901 compared to Investigator's choice of therapy as the 2L+ treatment for participants with advanced or metastatic gastric or GEJ adenocarcinoma expressing CLDN18.2, and the clinical performance of the investigational IVD. As part of this combined approach, the efficacy analyses from this study will also provide the basis to evaluate the clinical performance of Ventana CLDN18.2 assay as an IVD device for the identification of patients with advanced or metastatic gastric or GEJ adenocarcinoma expressing CLDN18.2 who may benefit from AZD0901.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent prior to any study procedure.
2. Participant must be at least 18 years or the legal age of consent in the jurisdiction in which the study is taking place at the time of signing the ICF.
3. Histologically confirmed unresectable, locally advanced or metastatic adenocarcinoma of gastric, GEJ, or distal esophagus (distal third of the esophagus) and the following requirement:

   (a) Participants with positive CLDN18.2 expression from archival tumor collected within past 24 months or from a fresh biopsy.
4. Disease progression on or after at least one prior line of treatment (LoT) for advanced or metastatic disease, which included a fluoropyrimidine and a platinum, for advanced or metastatic disease.
5. Must have at least one measurable or evaluable lesion assessed by the Investigator based on RECIST 1.1.
6. ECOG performance status of 0 or 1 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.
7. Predicted life expectancy of ≥ 12 weeks.
8. Adequate organ and bone marrow function
9. Body weight of ≥ 35 kg.
10. Sex and Contraceptive Requirements

Exclusion Criteria:

1. Participants with known HER2 positive status as defined as IHC 3+ or IHC 2+/ISH + (Cases with HER2: CEP17 ratio ≥ 2 or an average HER2 copy number ≥ 6.0 signals/cell are considered positive by ISH). Participants must undergo local (or have had) HER2 testing by IHC/ISH, and the most recent result of HER2 status will be used to determine the eligibility.
2. Participant has significant or unstable gastric bleeding and/or untreated gastric ulcers.
3. CNS metastases or CNS pathology including: epilepsy, seizures or aphasia within 3 months prior to consent, severe brain injury, dementia, Parkinson's disease, neurodegenerative diseases, cerebellar disease, severe uncontrolled mental illness, psychosis, CNS involvement of autoimmune diseases.
4. Participant has known clinically significant corneal disease (eg, active keratitis or corneal ulcerations).
5. Persistent toxicities (CTCAE Grade ≥ 2) caused by previous anticancer therapy, excluding alopecia. Participants with irreversible toxicity that is not reasonably expected to be exacerbated by study intervention may be included (eg, hearing loss).
6. Prior exposure to any ADC with MMAE payload or any CLDN18.2 targeting treatment other than naked monoclonal antibody (eg, CLDN18.2 targeting CAR-T cell therapy, multi-specific antibody including targeting CLDN18.2, etc).
7. History of thromboembolic events:

   1. Participants with venous thromboembolism within the past 6 months prior to randomization: participants with venous port or catheter thrombosis or superficial venous thrombus that do not require treatment or are stable on treatment with anticoagulants are excepted
   2. History of arterial thromboembolism within the past 12 months prior to randomization
8. As judged by the Investigator, any evidence of diseases which in the Investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardize compliance with the protocol.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-09-14 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in all randomized participants | From date of first dose/randomisation until disease progression or death in the absence of progression (approximately 3 years).
  The analysis will include all randomized participants. All events will be included, regardless of whether the participant withdraws from therapy or receives another anticancer therapy.
Overall Survival (OS) for 3L+ participants | From date of first dose/randomisation until the date of death due to any cause (approximately 3 years).
  The analysis will include all randomized participants who had at least 2 prior lines of systemic therapy. All deaths will be included, regardless of whether the participant withdraws from therapy or receives another anticancer therapy.

SECONDARY OUTCOMES:
OS in all randomized participants | From date of first dose/randomisation until the date of death due to any cause (approximately 3 years).
  The analysis will include all randomized participants. All deaths will be included, regardless of whether the participant withdraws from therapy or receives another anticancer therapy.
PFS for 3L+ participants | From date of first dose/randomisation until disease progression or death in the absence of progression (approximately 3 years).
  The analysis will include all randomized participants who had at least 2 prior lines of systemic therapy. All events will be included, regardless of whether the participant withdraws from therapy or receives another anticancer therapy.
Objective Response Rate (ORR) in all randomized participants | From date of first dose of AZD0901 up until progression, or the last evaluable assessment in the absence of progression (approximately 3 years).
  ORR is defined as the proportion of participants with at least one visit response of confirmed CR or confirmed PR, as determined by BICR per RECIST 1.1.
ORR for 3L+ participants | From date of first dose of AZD0901 up until progression, or the last evaluable assessment in the absence of progression (approximately 3 years).
  The analysis will include all randomized participants who had at least 2 prior lines of systemic therapy, with measurable disease at baseline
Duration of Response (DoR) in all randomized participants | From the date of first documented confirmed response until date of documented progression (approximately 3 years).
  The analysis will include all randomized participants with measurable disease at baseline who have a confirmed response. All events after achieving confirmed response will be included, regardless of whether the participant withdraws from therapy, receives another anticancer therapy or clinically progresses prior to RECIST 1.1.
Serum concentrations of AZD0901, total antibody and MMAE | From date of first dose of AZD0901 up until 30 days post AZD0901 discontinuation.
  To characterise the PK of AZD0901 in participants.
Status of ADA to AZD0901 | From date of first dose of AZD0901 up until 30 days post AZD0901 discontinuation.
  To determine the immunogenicity of AZD0901 in participants.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]. Changes from baseline in vital signs, clinical laboratory results, and ECGs | From start through 30 days post treatment completion and follow up for 90 days.
  To assess the safety and tolerability of AZD0901 as compared with Investigator's choice of therapy in all randomized participants who have received at least one dose of study intervention
PK parameters (such as peak concentration, as data allow) of AZD0901, total antibody and MMAE | From date of first dose of AZD0901 up until 30 days post AZD0901 discontinuation.
  To characterise the PK of AZD0901 in participants.
PK parameters (such as trough concentration, as data allow) of AZD0901, total antibody and MMAE | From date of first dose of AZD0901 up until 30 days post AZD0901 discontinuation.
  To characterise the PK of AZD0901 in participants.
Prevalence and incidence of ADA to AZD0901 | From date of first dose of AZD0901 up until 30 days post AZD0901 discontinuation.
  To determine the immunogenicity of AZD0901 in participants.
Titer of ADA to AZD0901 | From date of first dose of AZD0901 up until 30 days post AZD0901 discontinuation.
  To determine the immunogenicity of AZD0901 in participants.

CONTACTS AND LOCATIONS:
Locations (154):
- United States (33):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Duarte, California
  - Research Site, Fullerton, California
  - Research Site, Irvine, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Santa Rosa, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fleming Island, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Boise, Idaho
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Charlottesville, Virginia
  - Research Site, Fredericksburg, Virginia
  - Research Site, Olympia, Washington
  - Research Site, Seattle, Washington
- Brazil (4):
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
  - Research Site, Vitória
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Barrie, Ontario
  - Research Site, London, Ontario
  - Research Site, North York, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (26):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Lanzhou
  - Research Site, Lishui
  - Research Site, Luoyang
  - Research Site, Nanjing
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
- France (7):
  - Research Site, Besançon
  - Research Site, Brest
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Poitiers
- Germany (13):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, Moers
  - Research Site, München
- Research Site, Hong Kong, Hong Kong
- India (5):
  - Research Site, Ahmedabad
  - Research Site, Bengaluru
  - Research Site, Hyderabad
  - Research Site, Mumbai
  - Research Site, New Delhi
- Italy (7):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, Vicenza
- Japan (10):
  - Research Site, Fukuoka
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Ogaki-shi
  - Research Site, Osaka
  - Research Site, Sunto-gun
  - Research Site, Tokyo
  - Research Site, Toyoake-shi
  - Research Site, Yokohama
- Poland (9):
  - Research Site, Bielsko-Biala
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Szczecin
  - Research Site, Słupsk
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
- South Korea (2):
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Ourense
  - Research Site, Santander
  - Research Site, Seville
- Switzerland (4):
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Zurich
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Dusit
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Diyarbakır
  - Research Site, Erzurum
  - Research Site, Istanbul
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Taunton
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Vinh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Xu G, Liu W, Wang Y, Wei X, Liu F, He Y, Zhang L, Song Q, Li Z, Wang C, Xu R, Chen B. CMG901, a Claudin18.2-specific antibody-drug conjugate, for the treatment of solid tumors. Cell Rep Med. 2024 Sep 17;5(9):101710. doi: 10.1016/j.xcrm.2024.101710. Epub 2024 Sep 3. PMID 39232496